CLINICAL TRIAL: NCT03340038
Title: Use of a Non-ICU Specialty Ward For Immediate Post-operative Management of Head and Neck Free Flaps: A Randomized Controlled Trial
Brief Title: Use of a Non-ICU Specialty Ward For Immediate Post-operative Management of Head and Neck Free Flaps
Acronym: ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Arnaud Bewley, Assistant Professor Co-Director of Head and Neck Surgery Fellowship Director of Microvascular Reconstruction, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 841511
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Head and Neck Carcinoma; Trauma
Keywords: Free Flap Reconstructive Surgery; Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specialty Ward (Active Comparator): Patients who have been randomized into receiving post-operative care at the Non-ICU Specialty ward (intervention) after receiving flap reconstructive surgery on their mucosal or cutaneous defect.
  Interventions: Other: Non-ICU Specialty ward
- Intensive Care Unit (ICU) (No Intervention): Patients who have been randomized into receiving post-operative care at the intensive care unit after receiving flap reconstructive surgery on their mucosal or cutaneous defect.

INTERVENTIONS:
Other: Non-ICU Specialty ward
  Arms: Specialty Ward

SUMMARY:
Patients undergoing free flap reconstructive surgery at University of California, Davis Medical Center (UCDMC) will be assigned randomly into no intervention group (immediate post operative care in an ICU) or intervention group (immediate post operative care in a non-ICU specialty ward). The investigators hypothesize that there is no significant difference in the length of stay (LOS) or complication rate between head and neck free flaps patients managed immediately post-operatively in an ICU versus a non-ICU specialty ward. The primary objective is to compare the postoperative LOS between head and neck free-flap patients managed initially in an ICU versus a non-ICU specialty ward. The secondary objective is to compare differences in the rate of complications between head and neck free flap patients managed initially in an ICU versus a non-ICU specialty ward. Finally, the tertiary objective is to compare differences in resource utilization between head and neck free-flap patients managed initially in an ICU versus a non-ICU specialty ward.

DETAILED DESCRIPTION:
Free flaps are an instrumental component of head and neck reconstructive surgery. There is no current consensus on the postoperative management of these patients despite the increasing frequency with which free flaps are used. Although patients often do not have a specific medical indication for postoperative ICU management, they frequently are sent to the ICU for postoperative care based on the need for close nurse monitoring of the flap. In a US based survey in 2007, 88.9% of head and neck surgeons were sending postoperative flap patients to the ICU. Typical ICU length of stay for these patients varies from 2-11 days. There are numerous theoretic disadvantages to ICU care in these patients. ICU care has been associated with increased use of sedation leading to decreased flap perfusion, prolonged use of ventilation, less self care, less ambulation, increased delirium and increased cost.

Due to these concerns, several institutions have developed protocols that allow for the monitoring of head and neck free-flap patients outside of the ICU. Two recent retrospective studies assessed outcomes using these protocols, including 257 patients (119 ICU, 138 ward) and showed no significant difference in morbidity and mortality, or flap failure between the groups. There was a significant increase LOS from 8 to 9 days and transfusion rate, in the ICU group. Another study looked at 247 patients (175 ICU, 72 ward) and found no difference between flap failure, reoperation, hematoma, wound complications between the groups. They also found an increased LOS from 7 to 8 days in the ICU group. They calculated cost difference and found a decrease in average patient cost from $101,199 to $86,195 in the ward group. These studies support the use of non-ICU care for head and neck free-flap patients, however given their retrospective nature significant biases may exist, tempering the strength of their conclusions. To date, there has never been a Randomized Controlled Trial (RCT) that addresses this question.

This is a non-inferiority RCT at UCDMC to assess differences in LOS, complication rate and resource utilization between patients randomized to the ICU and a head and neck specialty ward. Since ICU/Ward bed availability has to be determined before surgery, a subject will be randomized before surgery when the subject meets all inclusion and none of the exclusion criteria. Currently, postoperative flap patients who are not enrolled in the study at UCDMC are monitored in the ICU for a minimum of 24 hours following their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing free flaps for reconstruction of head and neck surgical defects at UCDMC, including but not limited to, head and neck cancer defects, osteoradionecrosis (ORN), and trauma
* 18 years of age and older and able to consent

Exclusion Criteria:

* Vulnerable populations: adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-04-10 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Length of Stay | 30 days
  Number of days

SECONDARY OUTCOMES:
Inpatient Hospital Costs (dollar amounts) | 30 days
  Total inpatient hospital cost, insurance adjustments, and payments

OTHER OUTCOMES:
Post Operative Complication Rate | 30 days
  Flap ischemia, Reopration, Hematoma, wound infection, flap loss, and other complications
Medical Complications | 30 days
  Pneumonia, thromboembolic event, sepsis, ventilator requirement, cardiovascular complication, poster operative transfusion, delirium, ICU admission, other complications, mortality, readmission status

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bewley, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States